CLINICAL TRIAL: NCT06946979
Title: Clinical Study on the Use of Massage to Reconstruct the Function of Lumbar Stabilizer Muscles and Improve the "Muscle and Bone Imbalance" of Lumbar Disc Herniation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KLS-685-02
Record Dates: First submitted 2025-04-09; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Manipulation, Spinal; Dosage Forms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control group. (No Intervention)
- Spinal Manipulation + Medication Group. (Experimental): Spinal Manipulation Therapy :
  The treatment consists of two standardized steps: tendon adjustment techniques and bone-setting techniques.
  The total duration for both steps is approximately 15 minutes, conducted three times per week for two consecutive weeks.
  Pharmacotherapy :
  Patients in both groups will receive celecoxib (one tablet, twice daily) for two weeks, with detailed records maintained.
  Interventions: Other: Spinal Manipulation; Other: Medication
- Medication Group. (Active Comparator): Pharmacotherapy :
  Patients in both groups will receive celecoxib (one tablet, twice daily) for two weeks, with detailed records maintained.
  Interventions: Other: Medication

INTERVENTIONS:
Other: Spinal Manipulation — Spinal Manipulation Therapy The treatment consists of two standardized steps: tendon adjustment techniques and bone-setting techniques.
  The total duration for both steps is approximately 15 minutes, conducted three times per week for two consecutive weeks.
  Arms: Spinal Manipulation + Medication Group.
Other: Medication — Patients in both groups will receive celecoxib (one tablet, twice daily) for two weeks, with detailed records maintained.
  Arms: Medication Group.; Spinal Manipulation + Medication Group.

SUMMARY:
1. .Characterization of Stabilizing Muscle Dysfunction in LDH Patients Using advanced techniques such as high-density surface electromyography (HD-sEMG), this study will investigate the functional imbalance of lumbar stabilizing muscles in LDH patients by comparing their muscle function indicators to those of healthy controls.
2. .Impact of Spinal Manipulation on Lumbar Stabilizing Muscle Function Through serial sEMG evaluations, the study will assess changes in stabilizing muscle function in LDH patients before and after spinal manipulation. This includes a focus on endurance, motor control, and reaction time, providing evidence to inform the application of spinal manipulation in LDH treatment.
3. .Exploration of Mechanisms Underlying Spinal Manipulation in Improving "Musculoskeletal Imbalance" The study will examine correlations between improvements in stabilizing muscle function and clinical symptoms, such as pain relief and functional recovery. Statistical analyses of sEMG data and clinical efficacy indicators will be conducted to uncover the therapeutic characteristics of spinal manipulation in LDH intervention, offering new theoretical bases and strategies for long-term treatment and recurrence prevention.

ELIGIBILITY:
Inclusion Criteria:

* 1.Meet the diagnostic criteria for LDH as outlined in the ninth edition of "Surgery," with confirmation via MRI;
* 2.Age between 20 and 50;
* 3.Simple L4/5 disc herniation; VAS score ≥30/100;
* 4.Lumbar ODI index ≥20;
* 5.No massage, acupuncture, or physical therapy within the past month;
* 6.Signed informed consent form.

Exclusion Criteria:

* 1: Exclusion criteria: history of spinal surgery or severe spinal trauma;
* 2: combined with bone tuberculosis, tumors, severe osteoporosis, etc;
* 3: combined with serious internal diseases such as cardiovascular, hematological, digestive system diseases, or psychiatric disorders;
* 4: pregnant or lactating women;
* 5: combined with autoimmune diseases, allergic diseases, acute or chronic infectious diseases accompanied by pain and joint dysfunction;
* 6: MRI showing free nucleus pulposus or accompanied by cauda equina syndrome.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Lumbar Stabilizer Muscle Function Indicators. | week 3 (after the completion of the 2-week treatment period)
  Procedure: Patients lie prone on a table with the anterior superior iliac spine at the table edge. The upper body is suspended horizontally, arms crossed over the chest or extended parallel to the floor. Patients will maintain this posture for 90-120 seconds or until unable to continue (trunk angle deviation > 5°-10°). Surface electromyography (sEMG) signals will be collected synchronously, with three repetitions averaged.
  Electrode Placement: Surface EMG (ME6000, Finland) will be used to collect sEMG signals. Electrodes (0.5 cm diameter, 2 cm spacing) will be placed at the L5-S1 level for multifidus (LM) and L4-L5 for erector spinae (LE) muscles. Reference electrodes will be positioned 3 cm laterally. Sampling rate is set at 1000 Hz, with a bandpass filter of 10-500 Hz and noise level < 3.5 μV.
  Evaluation Metrics: Time-domain features and frequency-domain characteristics will be combined to report surface electromyography (sEMG) signals.

SECONDARY OUTCOMES:
Clinical efficacy indicators. | week 3 (after the completion of the 2-week treatment period)
  Pain will be assessed using the Visual Analogue Scale (VAS) , internationally recognized metrics for evaluating clinical efficacy in pain . Measurements will be conducted pre-treatment and after two weeks of intervention.
Clinical efficacy indicators. | week 3 (after the completion of the 2-week treatment period)
  Functional recovery will be assessed using theOswestry Disability Index (ODI), internationally recognized metrics for evaluating clinical efficacy in lumbar function. Measurements will be conducted pre-treatment and after two weeks of intervention.

IPD SHARING:
Plan to Share IPD: No